CLINICAL TRIAL: NCT02383524
Title: Does the Brain-derived Neurotrophic Factor Val66Met Gene Polymorphism Predict Inter-individual Variation in Responsiveness Following Lumbar Radiofrequency Denervation? A Single-centre, Prospective, Exploratory Study in Subjects Diagnosed With Zygapophysial Joint Pain
Brief Title: Genetic Predictors of Responsiveness to Radiofrequency Denervation in Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Parma (Other)
Responsible Party: Sponsor
Other Study IDs: 418120
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Low Back Pain (Lumbar Facet Joints Mediated Pain)
  Interventions: Procedure: Lumbar Radiofrequency Medial Branch Neurolysis

INTERVENTIONS:
Procedure: Lumbar Radiofrequency Medial Branch Neurolysis — Numerous studies have concluded that facet joint pain can be accurately diagnosed if a significant (but temporary) reduction in pain is achieved with a procedure called a Medial Branch Block (MBB). The clinician delivers a targeted injection of local anesthetic to the joint itself, or in close proximity to the medial branch of the posterior rami of the dorsal root. A significant decrease in pain confirms that the pain originates from the facet joint. If or when the pain returns after successful MBB treatment the patient may be considered for radiofrequency denervation (neurotomy) which selectively disrupts the joint's nerve supply and provides longer-term sustained relief

SUMMARY:
The Investigators have designed this exploratory study in patients suffering from zygapophysial joint mediated pain to investigate if a correlation exists between inter-individual genetic variability (genotype) with treatment response (phenotype). More specifically, the investigators aim to identify any form of correlation between a specific SNP of the BDNF gene (Val66Met) and the effectiveness and/or duration of radiofrequency facet joint neurotomy. The study population is patients suffering from chronic low back pain who have been scheduled for radiofrequency neurotomy following the diagnosis of facet joint mediated pain (using medial branch block test). The investigators will evaluate if a common variant of BDNF gene (Val66Met) can be directly correlated to a significant degree of pain relief following RF treatment, and whether the result of such a procedure can be predicted from a specific genetic profile.

DETAILED DESCRIPTION:
Study Hypothesis It is possible to predict individual responsiveness to radiofrequency denervation for zygapophysial (facet) joint mediated pain on the basis of a specific genetic pattern (Single Nucleotide Polymorphism, [SNP])?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic low back pain which is unresponsive to conservative treatment (including suitable analgesics and physical therapy);
* Willing to provide consent
* Subject is capable of comprehending the patient information sheet and has the capacity to give their informed consent to all study procedures in English
* Be 18 years or older at the time of enrolment;
* Have specific low back pain that is aggravated by hyperextension and rotation of the spine, with or without hip, buttock or leg pain that does not follow a known dermatomal distribution
* Paraspinal Tenderness
* A "positive" response to a uni/bi-lateral MBB* (a response is considered positive when a subject experiences at least 50% reduction in pain scores after the block, regardless of the duration of pain relief)

Exclusion Criteria:

* Patients who had had any previous back surgery
* Patients who had previous RF treatments for facet joints mediated pain
* Patients with another significant cause of low back pain (like spinal stenosis, disc herniation, spondylolisthesis, malignancy, infection or trauma);
* Radicular pain (pain with neuropathic characteristics following one or more nerve root distribution)
* Patients with bleeding complications or coagulopathy issues;
* Concurrent participation in other experimental trials;
* Known history of adverse reactions to local anesthetics;
* Pregnant or lactating women;
* Refusal to provide informed consent for blood banking
* Any other complication which in the view of the investigator may interfere with the study procedures or the measurement of the accurate study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic and debilitating low back pain with a diagnosis of lumbar zygapophysial joint mediated pain which has not been effectively treated with conservative pharmacological treatment or alternative non-invasive treatments
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Responder Rate | 3 months
  Number of patients in each group who report 50% reduction in pain on the visual analogue scale 3 months after radiofrequency denervation for lumbar zygapophysial (facet) joint mediated pain

SECONDARY OUTCOMES:
Medication intake, Functional status, Ability to work and Quality of life | 3 months

OTHER OUTCOMES:
Pre-specified Single Nucleotide Polymorphism (SNP) analysis | 3 months
  To evaluate whether any specific and/or combination of SNPs observed could be related with the clinical outcomes measured in this study

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's & St Thomas NHS Trust, London, United Kingdom